CLINICAL TRIAL: NCT02535351
Title: Targeted Therapy With or Without Nephrectomy in Metastatic Renal Cell Carcinoma: Liquid Biopsy for Biomarkers Discovery
Acronym: TARIBO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrolment
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 75/15; 2015-002240-14 (EudraCT Number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-28 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma
Keywords: Clear cell Metastatic renal cell carcinoma; Cytoreductive nephrectomy; First line treatment
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: TKIs (Active Comparator): sunitinib 50 mg orally 4 weeks on/ 2 weeks off or pazopanib 800 mg orally continuously
  Interventions: Drug: sunitinib or pazopanib
- B: TKIs + Cytoreductive Nephrectomy (Experimental): Cytoreductive nephrectomy + sunitinib 50 mg orally 4 weeks on/ 2 weeks off or pazopanib 800 mg orally continuously
  Interventions: Drug: sunitinib or pazopanib; Procedure: Cytoreductive nephrectomy

INTERVENTIONS:
Drug: sunitinib or pazopanib — First-line treatment
  Other Names: sutent or votrient
Procedure: Cytoreductive nephrectomy — Cytoreductive nephrectomy and first-line treatment
  Arms: B: TKIs + Cytoreductive Nephrectomy

SUMMARY:
Two randomized trials in the cytokine era clearly showed that cytoreductive nephrectomy (CN) had a role in metastatic renal cell carcinoma (mRCC) increasing life expectancy. The survival benefit of tyrosine kinase inhibitors (TKIs) including first-line sunitinib and pazopanib in mRCC has been demonstrated, but the majority of patients enrolled in the pivotal phase III studies had undergone nephrectomy.

Therefore it is unknown if similar survival benefit could be achieved without CN with these new targeted agents.

At the same time there is a need to better understand mechanisms of primary and secondary resistance to TKIs in mRCC patients and to identify eighter prognostic and predictive biomarkers to better define risk factors and potentially druggable targets.

DETAILED DESCRIPTION:
Two randomized trials in the cytokine era clearly showed that CN had a role in mRCC increasing life expectancy. The survival benefit of TKIs including first-line sunitinib and pazopanib in mRCC has been demonstrated, but the majority of patients enrolled in the pivotal phase III studies had undergone nephrectomy.Therefore it is unknown if similar survival benefit could be achieved without CN with these new targeted agents.

At the same time there is a need to better understand mechanisms of primary and secondary resistance to TKIs in mRCC patients and to identify eighter prognostic and predictive biomarkers to better define risk factors and potentially druggable targets.

The hypothesis of this study is that CN followed by TKIs will improve overall survival (OS) when compared to TKIs alone in subjects with mRCC. Circulating blood biomarkers (CBBs) promise to become non-invasive real-time surrogates for tissue-based biomarkers. Circulating tumor cells (CTCs) shed from both primary tumors and metastases, and circulating tumor DNA (ctDNA) released into the bloodstream from dying tumor cells, are likely to capture the entire tumor heterogeneity providing a clear picture of the tumor genetic landscape. Moreover, CTCs fluctuations reflect and possibly anticipate treatment outcome. Through comparison of CBBs before and after disease becomes refractory to therapy, the investigators would be able to address challenging research questions regarding TKIs resistance mechanisms.

This study was designed to compare clinical benefit as measured by Overall Survival (OS), progression-free survival (PFS), overall response rate (ORR) and safety provided by CN followed by TKIs vs upfront TKIs in mRCC subjects.To prospectively collect blood samples from patients at commencement of TKIs therapy and on development of resistance, with the purpose of analyzing CTCs and ctDNA mutational profile to highlight mechanisms underlying TKIs resistance. The investigators additionally aim to assess the role of CTCs as prognostic and pharmacodynamic biomarkers and prospectively collect demographic and clinical outcome data so that molecular and pathological analyses can be measured against clinical endpoints.

Rationale for TKIs treatment choice:

Pazopanib and sunitinib were compared to each other as a therapy for previously untreated patients with mRCC within the phase 3 non inferiority COMPARZ trial which represented the first-ever head-to-head comparison of first-line treatments for mRCC. Overall, the median PFS and OS with pazopanib compared to sunitinib were statistically non-inferior, showing that both agents are active and provide similar high quality care. For this reason the TKI will be assigned based on patients characteristics according to the guidelines of every single institution involved in the study.

Statistical plan:

The sample size was calculated in order to compare 5-year OS between subjects randomized to receive CN followed by TKIs and subjects randomized to receive TKIs (main study endpoint). A total of 191 deaths will yield 80% power to detect a hazard ratio of 1.5 of TKIs vs. CN followed by TKIs with an overall type 1 error of 0.05 (two-sided log-rank test). Such a hazard ratio (HR) corresponds to an increase in the 5-year OS, from an anticipated value 10% for TKIs to 21.5% for CN followed by TKIs. The investigators estimate that approximately 270 patients (135 in each arm), recruited over 3 years and with a minimum follow up of 2 years, will be necessary to see the necessary number of deaths.

An interim analysis of OS based on O'Brien-Fleming stopping rules is planned at 96 deaths at approximately 34 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ECOG Performance Status 0-1
* Favorable or intermediate MSKCC or Heng risk score
* Biopsy (primary tumour or metastases) confirming the diagnosis of predominantly clear cell RCC
* Resectable asymptomatic in situ primary (asymptomatic primary is defined as the absence of symptoms which can be exclusively assigned to the primary tumor such as flank pain and/or gross hematuria necessitating blood transfusion.)
* Tumour suitable to nephrectomy in the opinion of the urologist. Patients with Inferior vena cava thrombosis can be included
* Documented metastatic disease (CT scan or MRI)
* Life expectancy > or = 24 weeks
* Up to three different metastatic sites
* ≥ 3 metastatic lesions
* Platelets > 100,000/ml
* Haemoglobin > 9.0 g/dl
* neutrophils >1,500/mm3
* Bilirubin < or = 2 mg/dl, except for patients affected by Gilbert's syndrome
* AST and ALT < or = 2.5 times the UNL
* Serum albumin > the LNL
* Patients of childbearing age should use contraceptive methods during the study

Exclusion Criteria:

* Prior surgery or systemic treatment for mRCC
* Bilateral RCC
* Brain and liver metastases
* Non-clear-cell histology
* Poor prognosis as defined by MSKCC or Heng criteria
* Documented widespread disease (> or =4 metastatic organ sites)
* Oligometastatic disease suitable of metastasectomy (<3 lesions confined at one organ site)
* Symptomatic primary tumour at presentation
* High surgical risk in the opinion of the urologist
* Patients with > 3 of the following surgical risk factors are not eligible:

  * Serum albumin CTCAE v 4.0 grade 2 or worse
  * Serum LDH > 1.5 times upper limit of normal
  * Symptoms at presentation due to metastases
  * Clinical stage T4 disease
  * History of malabsorption syndrome
* Pregnant or breastfeeding women
* Concomitant cardiac disorders: cardiac failure NYHA> 2; Acute coronary syndrome or myocardial infarction or severe or unstable angina within the last 6 months as well as uncontrolled hypertension (sistolic>160, diastolic>90), arrhytmia requiring treatment (except for beta blockers or digossin)
* Uncontrolled diabetes
* Deep phlebitis not treated with LMWH or arterial thrombosis within the last 6 months
* HIV infection
* Active infections (> Grade 2 NCI-CTC v.3.0)
* Other cancer within the previous 5 years (except for in situ skin carcinoma, superficial bladder Ta, Tis, T1 and carcinoma of the cervix or every cancer with curative treatment within 5 years)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival benefit of cytoreductive nephrectomy with TKIs vs upfront TKIs in subjects with mRCC | 5 years
  To compare clinical benefit, as measured by Overall Survival (OS), provided by CN followed by TKIs vs upfront TKIs in subjects with mRCC

SECONDARY OUTCOMES:
Progression-free survival (PFS) and response rate (RR) benefit of cytoreductive nephrectomy with TKIs vs upfront TKIs | Radiological assessment: every 12 weeks (±1 week) until Progressive disease (up to 12 months) or treatment discontinuation (up to 5 years)
  To compare clinical benefit, as measured by progression-free survival (PFS) and response rate (RR) provided by CN followed by TKIs vs upfront TKIs
Safety profile (Adverse events) | day 1, every cycle (6 weeks for patients treated with Sunitinib and 4 weeks for patients treated with Pazopanib) until treatment discontinuation (up to 5 years).
  Safety profile of cytoreductive nephrectomy with TKIs vs upfront TKIs. (according to Common Terminology Criteria for Adverse Events -CTCAE- v 4.03). All Adverse events will be reported according to National Cancer Institute Criteria. The incidence of adverse events will be summarized according to the primary system-organ class (SOC) and within the category defined in the CTCAE v4.03. The summaries will be overall (severity grades 1-4) and for grade ≥3 events and will also report the actions taken in terms of treatment discontinuation. Similar summaries will be made for serious adverse events. The safety set will be considered.

OTHER OUTCOMES:
CTCs count | at baseline, pre- and post-operatively (in patients undergoing CN), 24 weeks after randomization and at the time of Progressive Disease up to 5 years
  To explore the association between baseline CTCs count and OS or PFS
CTCs count | at baseline, pre- and post-operatively (in patients undergoing CN), 24 weeks after randomization and at the time of Progressive Disease up to 5 years
  To compare baseline CTCs count and CTCs at the time of RECIST 1.1 PD on TKIs therapy, with the aim of better understand progressive changes in the tumor as resistance develops

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Mi, Italy

REFERENCES:
- [Background] Flanigan RC, Yonover PM. The role of radical nephrectomy in metastatic renal cell carcinoma. Semin Urol Oncol. 2001 May;19(2):98-102. PMID 11354539
- [Background] Flanigan RC, Salmon SE, Blumenstein BA, Bearman SI, Roy V, McGrath PC, Caton JR Jr, Munshi N, Crawford ED. Nephrectomy followed by interferon alfa-2b compared with interferon alfa-2b alone for metastatic renal-cell cancer. N Engl J Med. 2001 Dec 6;345(23):1655-9. doi: 10.1056/NEJMoa003013. PMID 11759643
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Flanigan RC, Mickisch G, Sylvester R, Tangen C, Van Poppel H, Crawford ED. Cytoreductive nephrectomy in patients with metastatic renal cancer: a combined analysis. J Urol. 2004 Mar;171(3):1071-6. doi: 10.1097/01.ju.0000110610.61545.ae. PMID 14767273
- [Background] Motzer RJ, Hutson TE, Cella D, Reeves J, Hawkins R, Guo J, Nathan P, Staehler M, de Souza P, Merchan JR, Boleti E, Fife K, Jin J, Jones R, Uemura H, De Giorgi U, Harmenberg U, Wang J, Sternberg CN, Deen K, McCann L, Hackshaw MD, Crescenzo R, Pandite LN, Choueiri TK. Pazopanib versus sunitinib in metastatic renal-cell carcinoma. N Engl J Med. 2013 Aug 22;369(8):722-31. doi: 10.1056/NEJMoa1303989. PMID 23964934
- [Background] Choueiri TK, Xie W, Kollmannsberger C, North S, Knox JJ, Lampard JG, McDermott DF, Rini BI, Heng DY. The impact of cytoreductive nephrectomy on survival of patients with metastatic renal cell carcinoma receiving vascular endothelial growth factor targeted therapy. J Urol. 2011 Jan;185(1):60-6. doi: 10.1016/j.juro.2010.09.012. Epub 2010 Nov 12. PMID 21074201
- [Background] Gossage L, Murtaza M, Slatter AF, Lichtenstein CP, Warren A, Haynes B, Marass F, Roberts I, Shanahan SJ, Claas A, Dunham A, May AP, Rosenfeld N, Forshew T, Eisen T. Clinical and pathological impact of VHL, PBRM1, BAP1, SETD2, KDM6A, and JARID1c in clear cell renal cell carcinoma. Genes Chromosomes Cancer. 2014 Jan;53(1):38-51. doi: 10.1002/gcc.22116. Epub 2013 Oct 29. PMID 24166983
- [Background] Heng DY, Wells JC, Rini BI, Beuselinck B, Lee JL, Knox JJ, Bjarnason GA, Pal SK, Kollmannsberger CK, Yuasa T, Srinivas S, Donskov F, Bamias A, Wood LA, Ernst DS, Agarwal N, Vaishampayan UN, Rha SY, Kim JJ, Choueiri TK. Cytoreductive nephrectomy in patients with synchronous metastases from renal cell carcinoma: results from the International Metastatic Renal Cell Carcinoma Database Consortium. Eur Urol. 2014 Oct;66(4):704-10. doi: 10.1016/j.eururo.2014.05.034. Epub 2014 Jun 13. PMID 24931622
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306